CLINICAL TRIAL: NCT03333785
Title: Improving Cancer Care Together Through eOncoNote
Brief Title: Randomized Trial of eOncoNote
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Clinical Oncology Group (OCOG) (Other); Ottawa Regional Cancer Centre (Other)
Responsible Party: Principal Investigator, Eva Grunfeld, Director, Knowledge Translation Research (OICR); Giblon Professor and Vice-Chair Research (Department of Family & Community Medicine, University of Toronto), University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OHSN-REB#20170381-01H; 128272 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2017-09-25; First posted 2017-11-07 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Communication Research; Breast Cancer; Prostate Cancer; Colorectal Cancer; Lung Cancer; Program, Communication; Remote Consultation
Keywords: Primary Care; Oncology; Continuity of care; Integration of care; Communication
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Communication; Neoplasms

STUDY DESIGN:
Intervention Model Description: Improving Cancer Care Together through eOncoNote is a concurrent mixed-methods hybrid type I effectiveness-implementation study design. Effectiveness of eOncoNote will be assessed by a pragmatic randomized controlled trial with individual patient randomization and outcomes measured at the patient level. Implementation will be assessed using a mixed methods process evaluation involving key stakeholders to assess barriers and facilitators to implementation of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Primary care providers whose patients have been randomized to the intervention group will receive an invitation from their patient's cancer specialist provider to communicate using eOncoNote. Primary care providers and cancer specialist providers will use eOncoNote in addition to usual methods of communication.
  Interventions: Behavioral: eOncoNote
- Control group (No Intervention): Primary care providers whose patients have been randomized to the control group will receive usual care (i.e. their primary care providers will not access eOncoNote to communicate with the cancer specialist providers and vice versa) and will be able to contact each other via telephone, fax, and mail consultation letters and progress notes, as per usual care.

INTERVENTIONS:
Behavioral: eOncoNote — * Diagnosis phase: The patient's nurse navigator will initiate an eOncoNote to the patient's PCP, inviting them to send any questions related to the patient's diagnostic process. The nurse navigator will initiate case closure after the diagnostic process has been completed (case will be open up to 4 months).
  * Treatment phase: The patient's medical or radiation oncologist will initiate an eOncoNote to the patient's PCP inviting them to ask questions related to the patient's cancer treatment and/or request information related to the patient's co-morbidities. The oncologist will initiate case closure after the treatment has been completed.
  * Survivorship phase: The patient's registered nurse within the Wellness Beyond Cancer Program will send an eOncoNote invitation to the patient's PCP inviting them to ask any questions as the patient transitions back to their care. The nurse will initiate case closure after one year.
  Arms: Intervention group

SUMMARY:
Improving Cancer Care Together through eOncoNote is a pragmatic randomized trial involving a secure online eConsultation system (referred to as eOncoNote) that will allow primary care providers and cancer specialist providers to communicate about their patients.

DETAILED DESCRIPTION:
The overall objectives of this randomized trial are to test an intervention designed to improve coordination/continuity of care between primary care providers (PCPs) and cancer specialist providers (CSPs), and to improve patient experience with regards to patients' perceived continuity of care. Participants will be patients at The Ottawa Hospital Cancer Centre in any one of three phases of the cancer continuum: diagnosis (colorectal, prostate, or lung cancer), active treatment (breast or prostate cancer) or survivorship (breast or colorectal cancer). The intervention involves a secure online eConsultation system that will allow PCPs and CSPs to communicate about their patient. Patients will be randomly allocated to one of two groups: 1) intervention group whereby their PCP and CSP will use a cancer-specific modification of the eConsultation system (eOncoNote) in addition to usual methods of communication or 2) control group receiving usual care (i.e. usual methods of communication such as telephone, fax, mailed consultation letters and progress notes). Randomization and outcomes will be at the level of the individual patient. The primary outcome is patients' perception of team/cross-boundary continuity. Secondary outcomes include measures of patients' anxiety and depression, and patients' experience of the care process. Qualitative methods including interviews with patients, PCPs, CSPs, and cancer system managers will also be conducted.

ELIGIBILITY:
Patient inclusion criteria:

* at least 18 years of age,
* being in one of the following three cancer continuum specific phases:

  1. Diagnosis phase: patients referred to the Cancer Assessment Clinic with suspected colorectal, prostate, or lung cancer;
  2. Treatment phase: patients receiving adjuvant chemotherapy for early stage breast cancer, or radical or adjuvant radiation therapy for localized prostate cancer;
  3. Survivorship phase: patients referred to the Wellness Beyond Cancer Program post completion of their adjuvant therapy for either breast or colorectal cancer with the intent of being discharged for survivorship care to their own family physician;
* no prior history of cancer in the past 5 years (those with non-melanoma skin cancer can participate).

Patient exclusion criteria:

* Currently participating in another study requiring ongoing completion of patient reported outcome measures (such as quality of life measures) in order to minimize respondent burden,
* Does not have a primary care provider,
* Patients will be excluded if their primary care provider has another patient enrolled in the trial in order to control for contamination between randomization groups,
* Inability to read and write in English,
* Inability to provide informed consent, and
* In the survivorship phase, patients who are discharged to the Wellness Beyond Cancer Program nurse practitioner (rather than their primary care providers) will be excluded.

Primary care providers eligibility criteria:

* Licensed family physician or nurse practitioner,
* Their patient has consented to be enrolled in the study, and they do not have any other patients enrolled in the study (to avoid contamination between intervention and control groups),
* They are already registered on the Champlain BASE(TM) eConsult system prior to their patient being enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Team/Cross Boundary Continuity subscale of the Nijmegen Continuity Questionnaire | Follow-up 2 = Diagnosis: 2 weeks; Treatment: 4 months for prostate cancer patients, 6 months for breast cancer patients; Survivorship: 12 months
  4-item subscale (scored on a five-point scale ranging from 1 = strongly disagree to 5 = strongly agree); calculate the mean of the items in the subscale

SECONDARY OUTCOMES:
Anxiety | (Follow-up 1 = Treatment: 1 month; Survivorship: 6 months); (Follow-up 2 = Diagnosis: 2 weeks; Treatment: 4 months for prostate cancer patients, 6 months for breast cancer patients; Survivorship: 12 months)
  Generalized Anxiety Disorder Screener (GAD-7); 7 items; 4 response options ("not at all" = 0; "several days" = 1; "more than half the days" = 2; "nearly every day" = 3)
Depression | (Follow-up 1 = Treatment: 1 month; Survivorship: 6 months); (Follow-up 2 = Diagnosis: 2 weeks; Treatment: 4 months for prostate cancer patients, 6 months for breast cancer patients; Survivorship: 12 months)
  Patient Health Questionnaire on major depression (PHQ-9); 10 items in total; items 1-9: 4 response options ("not at all" = 0; "several days" = 1; "more than half the days" = 2; "nearly every day" = 3); item 10: four-point scale (ranging from "not difficult at all" to "extremely difficult")
Patient experience of the care process | (Follow-up 1 = Treatment: 1 month; Survivorship: 6 months); (Follow-up 2 = Diagnosis: 2 weeks; Treatment: 4 months for prostate cancer patients, 6 months for breast cancer patients; Survivorship: 12 months)
  Picker Patient Experience Questionnaire (PPE-15); 15 items; each item scored as dichotomous score indicating presence or absence of a problem (defined as an aspect of health care that could be improved upon from the patient's perspective)

OTHER OUTCOMES:
Team/Cross Boundary Continuity subscale of the Nijmegen Continuity Questionnaire | Follow-up 1 = Treatment: 1 month; Survivorship: 6 months
  4-item subscale (scored on a five-point scale ranging from 1 = strongly disagree to 5 = strongly agree); calculate the mean of the items in the subscale

CONTACTS AND LOCATIONS:
Overall Officials: Eva Grunfeld, MD, DPhil, Principal Investigator — University of Toronto; Sharon McGee, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrovic B, Julian JA, Liddy C, Afkham A, McGee SF, Morgan SC, Segal R, Sussman J, Pond GR, O'Brien MA, Bender JL, Grunfeld E. Web-Based Asynchronous Tool to Facilitate Communication Between Primary Care Providers and Cancer Specialists: Pragmatic Randomized Controlled Trial. J Med Internet Res. 2023 Jan 18;25:e40725. doi: 10.2196/40725. PMID 36652284
- See also: Champlain BASE eConsult Website — http://www.champlainbaseeconsult.com/